CLINICAL TRIAL: NCT02929108
Title: ACCESS (Access for Cancer Caregivers for Education and Support for Shared Decision)
Brief Title: ACCESS (Access for Cancer Caregivers for Education and Support for Shared Decision Making)
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Debra Parker Oliver, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006270; 5R01CA203999 (NIH)
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Cancer; Pain
Keywords: hospice; caregiver
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: A pragmatic cluster randomized controlled trial will randomly assign hospice sites (cluster) to 2 of 3 groups: 1) Enhanced usual care 2) Enhanced usual care and private Facebook group 3) Enhanced usual care, private Facebook group, and ACCESS. Each hospice site (cluster) will go through 2 arms of the intervention but the family caregiver participants will only complete one arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Usual Care (No Intervention): The family caregivers in his group will receive usual hospice care which has been enhanced as the staff have been trained in shared decision making.
- Facebook (Experimental): The family caregivers in this group only participates in the Facebook groups, not in the shared decision making
  Interventions: Behavioral: Facebook
- ACCESS (Experimental): The family caregivers in this group participates in Facebook and web conferencing for shared decision making
  Interventions: Behavioral: Facebook; Behavioral: ACCESS

INTERVENTIONS:
Behavioral: Facebook — Participants will be enrolled in a Secret Facebook group for social support and education
  Arms: ACCESS; Facebook
Behavioral: ACCESS — Intervention will have two components.
  1. Participants will be enrolled in a Secret Facebook group for social support and education
  2. Participants will use web conferencing technology to participate in their interdisciplinary team meeting
  Arms: ACCESS

SUMMARY:
The project will test the effect of educating and supporting family caregivers of hospice cancer patients on their active participation in shared decision making in the plan of care for their patients.

DETAILED DESCRIPTION:
This intervention will target education and emotional support to family caregivers of hospice cancer patients for a shared decision making process in the hospice care plan meetings The intervention ACCESS will consist of three components:

1: a Facebook group to provide the education and support; 2. web conferencing for family members into the hospice interdisciplinary care plan meeting 3, a structured shared decision making process to guide the team discussion.

Participants (family caregivers) will be randomly assigned to one of three groups, usual care, Facebook only, and Access.

The specific aims are to:

1. Evaluate the effect of access on family caregiver anxiety, pain knowledge and patient pain.
2. Evaluate the effect of Facebook groups as educational emotional support for family caregivers
3. Assess staff and family caregiver satisfaction with the shared decision making process.

ELIGIBILITY:
Inclusion Criteria:

* Is caregiving for a patient enrolled in the participating hospice
* Over 18 years of age
* Is caregiving for a patient with a diagnosis of cancer
* Willing to have a Facebook account and post at least 1x per week if in intervention group

Exclusion Criteria:

* No one under the age of 18
* Is caregiving for a patient enrolled in hospice agencies other than those participating in the study
* Unwilling to participate in social media
* Is caregiving for a patient with a diagnosis other than cancer
* Is caregiving for a patient with a life expectancy of less than 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Oliver, PhD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Hospice Compassus, Columbia, Missouri
  - CrossRoads Hospice, Kansas City, Missouri
  - Barnes Jewish Hospice, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker Oliver D, Demiris G, Washington KT, Pitzer K, Ulrich C. The Effect of Digital Literacy on Participation in Social Media Clinical Trials in Cancer: Tailoring an Informed Consent Process. Telemed J E Health. 2022 Mar 21;28(11):1682-9. doi: 10.1089/tmj.2021.0555. Online ahead of print. PMID 35324322
- [Derived] Oliver DP, Washington KT, Pitzer K, Popejoy L, White P, Wallace AS, Grimsley A, Demiris G. Mixed methods analysis of hospice staff perceptions and shared decision making practices in hospice. Support Care Cancer. 2022 Mar;30(3):2679-2691. doi: 10.1007/s00520-021-06631-w. Epub 2021 Nov 25. PMID 34825279
- [Derived] Starr LT, Bullock K, Washington K, Aryal S, Parker Oliver D, Demiris G. Anxiety, Depression, Quality of Life, Caregiver Burden, and Perceptions of Caregiver-Centered Communication among Black and White Hospice Family Caregivers. J Palliat Med. 2022 Apr;25(4):596-605. doi: 10.1089/jpm.2021.0302. Epub 2021 Nov 18. PMID 34793244
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a crossover cluster-randomized study where 7 hospice sites were assigned to an intervention sequence consisting of 2 of the 3 interventions: Facebook, Enhanced UsualCare, or ACCESS. There was at least one washout period of up to 90 days between interventions. The intervention for the hospice sites also started at different times.
Pre-assignment Details: Hospice patients were not enrolled to this study. Only family caregivers were enrolled to this study. Each family caregiver was only assigned to one group (intervention) and stayed in that group for the duration of their time in the study (up to 90 days). They were given surveys at 14, 28, 60, and 90 days. The number of family caregivers who received each intervention at each site is listed below.
Groups:
- Site 1: Facebook First, Then Access, Then Facebook: This site was assigned to the intervention sequence: Facebook First, Then Access, Then Facebook, and started in August 2017. Each intervention was approximately 12 months in length, with up to a 3-month washout period between interventions. Caregivers only received one intervention for up to 90 days.
- Site 2: Access First Then Enhanced Usual Care, Then Access: This site was assigned to the intervention sequence: Access First, Then Enhanced Usual Care, Then Access, and started in November 2017. Each intervention was approximately 12 months in length, with up to a 3-month washout period only between the first and second intervention. Caregivers only received one intervention for up to 90 days.
- Site 3: Access First, Then Enhanced Usual Care, Then Access: This site was assigned to the intervention sequence: Access First, Then Enhanced Usual Care, Then Access, and started in December 2017. Each intervention was approximately 12 months in length, with up to a 3-month washout period only between the first and second intervention. Caregivers only received one intervention for up to 90 days.
- Site 4: Enhanced Usual Care First, Then Facebook, Then Enhanced Usual Care: This site was assigned to the intervention sequence: Enhanced Usual Care First, Then Facebook, Then Enhanced Usual Care, and started in December 2017. Each intervention was approximately 12 months in length, with up to a 3-month washout period only between the second and third intervention. Caregivers only received one intervention for up to 90 days.
- Site 5: Facebook First, Then Enhanced Usual Care, Then Facebook: This site was assigned to the intervention sequence: Access First, Then Enhanced Usual Care, Then Access, and started in January 2018. Each intervention was approximately 12 months in length, with up to a 3-month washout period only between the first and second intervention. Caregivers only received one intervention for up to 90 days.
- Site 6: Enhanced Usual Care First, Then Facebook, Then Enhanced Usual Care: This site was assigned to the intervention sequence: Enhanced Usual Care First, Then Facebook, Then Enhanced Usual Care, and started in February 2018. Each intervention was approximately 12 months in length, with up to a 3-month washout period only between the second and third intervention. Caregivers only received one intervention for up to 90 days.
- Site 7: Access First ,Then Facebook: This site was assigned to the intervention sequence: Access First, Then Facebook, and started in September 2019. Each intervention was approximately 12 months in length, with up to a 3-month washout period between both interventions. Caregivers only received one intervention for up to 90 days.
Period: Overall Study
Arm/Group | Site 1: Facebook First, Then Access, Then Facebook | Site 2: Access First Then Enhanced Usual Care, Then Access | Site 3: Access First, Then Enhanced Usual Care, Then Access | Site 4: Enhanced Usual Care First, Then Facebook, Then Enhanced Usual Care | Site 5: Facebook First, Then Enhanced Usual Care, Then Facebook | Site 6: Enhanced Usual Care First, Then Facebook, Then Enhanced Usual Care | Site 7: Access First ,Then Facebook
Started | 122 | 75 | 39 | 60 | 73 | 32 | 88
Facebook | 94 | 0 | 0 | 11 | 57 | 10 | 42
Access (Although the hospice site was assigned Facebook and Enhanced Usual Care, there were 5 caregivers that did receive the intervention of Access.) | 28 | 47 | 23 | 0 | 5 | 0 | 46
Enhanced Usual Care | 0 | 28 | 16 | 49 | 11 | 22 | 0
Completed | 22 | 11 | 11 | 14 | 18 | 4 | 10
Not Completed | 100 | 64 | 28 | 46 | 55 | 28 | 78
Not completed — Hospice patient death | 100 | 64 | 28 | 46 | 55 | 28 | 78

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Usual Care: The family caregivers in this group will receive usual hospice care which has been enhanced as the staff have been trained in shared decision making.
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care | Facebook | ACCESS | Total
Number analyzed (Participants) | 126 | 214 | 149 | 489
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age is missing for some participants.
  years
    number analyzed (Participants) | 125 | 214 | 143 | 482
    (all) | 57.8 (12.2) | 55.0 (12.8) | 56.5 (12.0) | 56.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex is missing for one participant.
  Participants
    number analyzed (Participants) | 126 | 214 | 148 | 488
    Female | 87 | 169 | 119 | 375
    Male | 39 | 45 | 29 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 4 | 10
  Not Hispanic or Latino | 125 | 209 | 141 | 475
  Unknown or Not Reported | 0 | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 34 | 16 | 56
  White | 118 | 172 | 125 | 415
  More than one race | 2 | 1 | 3 | 6
  Unknown or Not Reported | 0 | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 126 | 214 | 149 | 489

OUTCOME MEASURES:

1. Primary Outcome: Change in Generalized Anxiety Disorder- 7
Description: A screening tool to quantify participant's anxiety. The scale ranges from 0-21. A higher score indicates a higher level of anxiety.
Time Frame: Upon enrollment, 14 days, 28 days, 60 days and 90 days
Population: Some questionnaires were not completed by the participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Facebook | ACCESS
Number analyzed (Participants) | 126 | 214 | 149
score on a scale
  Baseline (upon enrollment): number analyzed (Participants) | 119 | 199 | 140
  Baseline (upon enrollment) | 7.73 (5.84) | 8.81 (5.98) | 8.42 (5.73)
  14 days: number analyzed (Participants) | 80 | 117 | 98
  14 days | 7.06 (5.97) | 6.93 (5.28) | 7.39 (5.03)
  28 days: number analyzed (Participants) | 52 | 90 | 53
  28 days | 6.81 (5.74) | 6.02 (4.50) | 7.55 (4.98)
  60 days: number analyzed (Participants) | 35 | 59 | 32
  60 days | 5.06 (4.82) | 6.54 (4.20) | 8.81 (5.69)
  90 days: number analyzed (Participants) | 30 | 40 | 23
  90 days | 6.43 (5.52) | 6.10 (3.91) | 7.43 (4.52)

2. Secondary Outcome: Change in Family Pain Questionnaire - Experience
Description: A scale which measures caregiver's experience dealing with patient pain. Scale ranges from 0-70. A higher score indicates higher pain experience.
Time Frame: Upon enrollment and 28 days
Population: Some questionnaires were not completed by the participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Facebook | ACCESS
Number analyzed (Participants) | 126 | 214 | 149
score on a scale
  Baseline (upon enrollment): number analyzed (Participants) | 113 | 184 | 136
  Baseline (upon enrollment) | 38.9 (11.0) | 40.9 (10.8) | 40.2 (11.0)
  28 days: number analyzed (Participants) | 32 | 49 | 38
  28 days | 39.3 (10.7) | 39.0 (9.53) | 40.8 (9.88)

3. Secondary Outcome: Change in Family Pain Questionnaire - Knowledge
Description: A scale which measures pain knowledge. The scale ranges from 0-90. A higher score indicates a higher knowledge of pain.
Time Frame: Upon enrollment and 28 days
Population: Some questionnaires were not completed by the participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Facebook | ACCESS
Number analyzed (Participants) | 126 | 214 | 149
score on a scale
  Baseline (upon enrollment): number analyzed (Participants) | 112 | 182 | 126
  Baseline (upon enrollment) | 53.2 (12.4) | 54.6 (11.2) | 54.3 (11.0)
  28 days: number analyzed (Participants) | 32 | 51 | 41
  28 days | 60.9 (11.3) | 55.2 (11.0) | 54.8 (8.75)

4. Secondary Outcome: Change in Caregiver Quality of Life
Description: Four question scale that measures caregivers quality of life. Scale ranges from 0-40. Higher score indicates higher quality of life.
Time Frame: Upon enrollment, 14 days, 28 days, 60 days and 90 days
Population: Some questionnaires were not completed by the participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Facebook | ACCESS
Number analyzed (Participants) | 126 | 214 | 149
score on a scale
  Baseline (upon enrollment): number analyzed (Participants) | 122 | 208 | 143
  Baseline (upon enrollment) | 26.7 (8.76) | 24.4 (8.26) | 24.9 (8.19)
  14 days: number analyzed (Participants) | 80 | 117 | 97
  14 days | 25.1 (9.33) | 24.8 (7.59) | 24.3 (7.60)
  28 days: number analyzed (Participants) | 52 | 90 | 53
  28 days | 25.3 (9.40) | 23.6 (7.92) | 22.6 (7.14)
  60 days: number analyzed (Participants) | 34 | 59 | 32
  60 days | 27.0 (8.12) | 22.6 (8.06) | 21.9 (8.57)
  90 days: number analyzed (Participants) | 30 | 39 | 22
  90 days | 26.3 (8.03) | 22.7 (6.91) | 23.4 (6.73)

5. Secondary Outcome: Perceived Involvement of Care Scale
Description: A scale measuring perceived involvement of care. Scale ranges from 13-65. Higher score indicates higher perceived involvement in care.
Time Frame: Upon enrollment, 14 days, 28 days, and 90 days
Population: Some questionnaires were not completed by the participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Facebook | ACCESS
Number analyzed (Participants) | 126 | 214 | 149
score on a scale
  Baseline (upon enrollment): number analyzed (Participants) | 74 | 125 | 121
  Baseline (upon enrollment) | 44.1 (8.69) | 43.7 (10.6) | 42.9 (8.85)
  14 days: number analyzed (Participants) | 33 | 45 | 15
  14 days | 41.0 (8.93) | 42.5 (9.35) | 43.9 (9.22)
  28 days: number analyzed (Participants) | 34 | 55 | 47
  28 days | 41.8 (10.8) | 44.3 (9.95) | 46.3 (6.24)
  90 days: number analyzed (Participants) | 23 | 19 | 18
  90 days | 45.4 (10.8) | 45.9 (8.58) | 49.3 (6.88)

6. Secondary Outcome: Public Health Questionnaire (PHQ 9)
Description: A measure of depression. Scale ranges from 0-27. A higher score indicates higher depression.
Time Frame: Upon enrollment, 14 days, 28 days, 60 days, and 90 days
Population: Some questionnaires were not completed by the participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Facebook | ACCESS
Number analyzed (Participants) | 126 | 214 | 149
score on a scale
  Baseline (upon enrollment): number analyzed (Participants) | 115 | 202 | 143
  Baseline (upon enrollment) | 7.05 (6.59) | 7.88 (6.20) | 7.87 (6.30)
  14 days: number analyzed (Participants) | 80 | 117 | 98
  14 days | 6.43 (6.37) | 6.30 (5.24) | 6.82 (5.41)
  28 days: number analyzed (Participants) | 52 | 90 | 53
  28 days | 6.37 (6.47) | 6.18 (4.86) | 6.85 (4.64)
  60 days: number analyzed (Participants) | 35 | 59 | 32
  60 days | 4.74 (5.24) | 6.20 (4.65) | 7.91 (5.84)
  90 days: number analyzed (Participants) | 30 | 39 | 23
  90 days | 5.50 (4.98) | 5.59 (4.04) | 6.43 (4.08)

7. Secondary Outcome: Edmonton Symptom Assessment
Description: A scale that measures various patient symptoms as reported by caregiver such as pain, fatigue, depression, anxiety, appetite, and nausea. Scale ranges from 0-90. A higher score indicates higher degree of symptoms.
Time Frame: Upon enrollment, 14 days, 28 days, 60 days, and 90 days
Population: Some questionnaires were not completed by the participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Facebook | ACCESS
Number analyzed (Participants) | 126 | 214 | 149
score on a scale
  Baseline (upon enrollment): number analyzed (Participants) | 51 | 73 | 27
  Baseline (upon enrollment) | 45.6 (15.9) | 46.1 (14.3) | 42.6 (13.5)
  14 days: number analyzed (Participants) | 80 | 114 | 96
  14 days | 43.6 (16.3) | 42.2 (15.1) | 43.6 (14.6)
  28 days: number analyzed (Participants) | 19 | 34 | 6
  28 days | 51.6 (17.7) | 41.7 (14.5) | 27.5 (10.3)
  60 days: number analyzed (Participants) | 34 | 59 | 32
  60 days | 43.9 (15.6) | 43.4 (15.2) | 45.4 (14.2)
  90 days: number analyzed (Participants) | 30 | 39 | 21
  90 days | 51.2 (17.6) | 42.3 (14.1) | 42.0 (16.7)

8. Secondary Outcome: Zarit Burden Scale
Description: A scale that measures the level of burden on caregiver. Scale ranges from 0-28. A higher score indicates greater burden.
Time Frame: Upon enrollment and 28 days
Population: Some questionnaires were not completed by the participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Facebook | ACCESS
Number analyzed (Participants) | 126 | 214 | 149
score on a scale
  Baseline (upon enrollment): number analyzed (Participants) | 120 | 205 | 145
  Baseline (upon enrollment) | 8.78 (6.05) | 9.74 (6.26) | 10.3 (6.25)
  28 days: number analyzed (Participants) | 53 | 90 | 53
  28 days | 9.53 (5.58) | 9.79 (4.82) | 10.7 (5.15)

9. Secondary Outcome: Caregiver Communication Questionnaire (CCCQ)
Description: A scale that measures the level of perception of caregiver centered communication by hospice staff. Scale ranges from 30-150. A higher score indicates greater perception of caregiver centered communication.
Time Frame: 14 days, 28 days, and 60 days
Population: Some questionnaires were not completed by the participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Facebook | ACCESS
Number analyzed (Participants) | 126 | 214 | 149
score on a scale
  14 days: number analyzed (Participants) | 80 | 112 | 95
  14 days | 117 (19.9) | 112 (22.5) | 117 (20.7)
  28 days: number analyzed (Participants) | 19 | 34 | 6
  28 days | 120 (26.9) | 119 (20.9) | 114 (24.0)
  60 days: number analyzed (Participants) | 26 | 32 | 28
  60 days | 116 (22.1) | 116 (21.0) | 121 (20.0)

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality was followed from baseline through completion of follow-up (up to 90 days).
Arm/Group | Enhanced Usual Care | Facebook | ACCESS
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/214 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/214 | 0/149
Other Adverse Events (participants affected / at risk) | 0/126 | 0/214 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT02929108/Prot_SAP_000.pdf